CLINICAL TRIAL: NCT05954767
Title: A Phase 3 Multi-Center Efficacy Study of IS-001 Injection in Patients Undergoing Robotic-Assisted Gynecological Surgery Using the da Vinci® Surgical System With Firefly® Fluorescent Imaging
Brief Title: IS-001 Injection in Patients Undergoing Robotic-Assisted Gynecological Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISI-124804-3
Record Dates: First submitted 2023-06-01; First posted 2023-07-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: Ureter Injury
MeSH Terms: interventions — IS 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efficacy (Other): Single intravenous injection of IS-001 and ureter visualization and delineation will be compared in white light standard of care and near-infrared (NIR) imaging mode.
  Interventions: Drug: IS-001

INTERVENTIONS:
Drug: IS-001 — IV injection of IS-001 drug substance with near infrared (NIR) imaging

SUMMARY:
This study evaluates the safety and efficacy of intravenous injection of IS-001 to aid in intraoperative ureter structure delineation.

DETAILED DESCRIPTION:
Injury to the ureter, the duct by which urine passes from the kidney into the bladder, is a well-known and serious complication of pelvic and abdominal surgery that frequently goes unrecognized intraoperatively. This study seeks to evaluate the safety and efficacy of intravenous IS-001 injection to improve surgeon ureter visualization during robotic-assisted surgery with the da Vinci® Surgical System and Firefly® imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject is between the ages of 16 and 75, inclusive at time of consent.
2. Subject is scheduled to undergo robotic-assisted gynecological procedure using a da Vinci® Surgical System with Firefly® Fluorescence Imaging.
3. Subject and/or subject's parent/guardian is willing and able to provide informed consent and/or assent as applicable.

Exclusion Criteria:

1. Subject is pregnant or nursing.
2. Subject has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
3. Subject is already enrolled in another investigational drug or device study receiving therapeutic agents within the past 6 months
4. Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete quality data or represents an unacceptable safety profile
5. Subject has a known or suspected hypersensitivity to indocyanine green (ICG)
6. Subject has any of the following screening laboratory values:

   1. eGFR < 60 mL/min/1.73 m^2
   2. Aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase (SGOT) ≥ 2.5 × ULN
   3. Alanine aminotransferase (ALT) or serum glutamic pyruvic transaminase (SGPT) ≥ 2.5 × ULN.
7. Planned use of CYTALUX™ (pafolacianine) for surgery

Ages: 16 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — biological
Enrollment: 189 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible. | 10 minutes
  Evaluate ureter visualization by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 10 minutes after IS-001 injection
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 30 minutes
  Evaluate ureter visualization by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 30 minutes after IS-001 injection

SECONDARY OUTCOMES:
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length | 10
  Evaluate ureter length delineation by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 10 minutes after injection
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length | 30
  Evaluate ureter length delineation by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 30 minutes after injection
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 10 minutes
  Evaluate ureter visualization based on intraoperative surgeon's rating at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 10 minutes after IS-001 injection
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 30 minutes
  Evaluate ureter visualization based on intraoperative surgeon's rating at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 30 minutes after IS-001 injection
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 45 minutes
  Evaluate ureter visualization by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 45 minutes after IS-001 injection
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length | 45 minutes
  Evaluate ureter length delineation by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 45 minutes after IS-001 injection
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible | 45 minutes
  Evaluate ureter visualization based on intraoperative surgeon's rating at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode at 45 minutes after IS-001 injection
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in near infrared imaging mode | 10 minutes
  Evaluate ureter signal-to-background ratio in Firefly imaging across time points at (a) the pelvic brim location and (b) the uterine arteries location after IS-001 injection.
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in near infrared imaging mode | 30 minutes
  Evaluate ureter signal-to-background ratio in Firefly imaging across time points at (a) the pelvic brim location and (b) the uterine arteries location after IS-001 injection.
Ureter signal-to-background ratio evaluating contrast of fluorescent signal in near infrared imaging mode | 45 minutes
  Evaluate ureter signal-to-background ratio in Firefly imaging across time points at (a) the pelvic brim location and (b) the uterine arteries location after IS-001 injection.
concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 10 minutes
  Determine degree of concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment at (a) the pelvic brim location and (b) the uterine arteries location
concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 30 minutes
  Determine degree of concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment at (a) the pelvic brim location and (b) the uterine arteries location
concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment | 45 minutes
  Determine degree of concordance between intra-operative ureter visualization assessment and independent reader ureter visualization assessment at (a) the pelvic brim location and (b) the uterine arteries location
Determine degree of concordance of ureter visualization between independent readers | 10 minutes
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim location and (b) the uterine arteries location
Determine degree of concordance of ureter visualization between independent readers | 30 minutes
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim location and (b) the uterine arteries location
Determine degree of concordance of ureter visualization between independent readers | 45 minutes
  Determine degree of concordance of ureter visualization between independent readers at (a) the pelvic brim location and (b) the uterine arteries location
degree of concordance of ureter visualization within independent readers | 10 minutes
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim location and (b) the uterine arteries location
degree of concordance of ureter visualization within independent readers | 30 minutes
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim location and (b) the uterine arteries location
degree of concordance of ureter visualization within independent readers | 45 minutes
  Determine degree of concordance of ureter visualization within independent readers at (a) the pelvic brim location and (b) the uterine arteries location

OTHER OUTCOMES:
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible after second injection | 10 minutes
  Evaluate ureter visualization by independent reader at (a) the pelvic brim and (b) uterine arteries in Firefly® imaging compared white light mode after 2nd IS-001 injection for procedures lasting longer than 60 minutes
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible after second injection | 30 minutes
  Evaluate ureter visualization by independent reader at (a) the pelvic brim and (b) uterine arteries in Firefly® imaging compared white light mode after 2nd IS-001 injection for procedures lasting longer than 60 minutes
Independent reader assessment of ureter visualization by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible after second injection | 45 minutes
  Evaluate ureter visualization by independent reader at (a) the pelvic brim and (b) uterine arteries in Firefly® imaging compared white light mode after 2nd IS-001 injection for procedures lasting longer than 60 minutes
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length after second injection | 10 minutes
  Evaluate ureter length delineation by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode after second injection for procedures lasting longer than 60 minutes
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length after second injection | 30 minutes
  Evaluate ureter length delineation by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode after second injection for procedures lasting longer than 60 minutes.
Independent reader assessment of ureter length delineation by line drawing on recorded frame measured in arbitrary unit length after second injection | 45 minutes
  Evaluate ureter length delineation by independent reader at (a) the pelvic brim and (b) uterine arteries location in Firefly® mode compared to white light mode after second injection for procedures lasting longer than 60 minutes.
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible - 2nd injection | 10 minutes
  Evaluate ureter visualization based on intraoperative surgeon's rating at (a) the pelvic brim and (b) uterine arteries in Firefly® imaging over white light mode after 2nd IS-001 injection for procedures lasting longer than 60 minutes
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible - 2nd injection | 30 minutes
  Evaluate ureter visualization based on intraoperative surgeon's rating at (a) the pelvic brim and (b) uterine arteries in Firefly® imaging over white light mode after 2nd IS-001 injection for procedures lasting longer than 60 minutes
Ureter visualization based on intraoperative surgeon's rating by 1-5 Likert visualization rating scale from 1 not visible, 2 questionably visible, 3 low visibility, 4 visible, 5 clearly visible - 2nd injection | 45 minutes
  Evaluate ureter visualization based on intraoperative surgeon's rating at (a) the pelvic brim and (b) uterine arteries in Firefly® imaging over white light mode after 2nd IS-001 injection for procedures lasting longer than 60 minutes

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - HCA Mercy Hospital, Miami, Florida
  - Orlando Health, Orlando, Florida
  - E.W. Sparrow Hospital, Lansing, Michigan
  - MountainView Hospital, Las Vegas, Nevada
  - The Ohio State Unversity, Columbus, Ohio
  - OhioHealth, Columbus, Ohio
  - St. David's Surgical Hospital, Austin, Texas